CLINICAL TRIAL: NCT03152643
Title: Cumulative Live Birth Rates After Cleavage-stage Versus Blastocyst-stage Embryo Transfer: A Multicenter, Prospective, Randomized Controlled Trial
Brief Title: Cumulative Live Birth Rates After Cleavage-stage Versus Blastocyst-stage Embryo Transfer
Acronym: CLBR-CBSET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Shandong Provincial Hospital (Other Government); RenJi Hospital (Other); Guangxi Maternal and Child Health Hospital (Other); Third Affiliated Hospital of Zhengzhou University (Other); Shengjing Hospital (Other); The Third Affiliated Hospital of Guangzhou Medical University (Other); General Hospital of Ningxia Medical University (Other); Suzhou Municipal Hospital (Other); Henan Provincial People's Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLBR-CBSET
Record Dates: First submitted 2017-05-09; First posted 2017-05-15 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Infertility
Keywords: Cumulative live birth rates; cleavage-stage embryo transfer; blastocyst transfer
MeSH Terms: conditions — Infertility | interventions — Embryo Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- blastocyst-stage embryo transfer group (Experimental): For subjects assigned to blastocyst-stage (D5/D6) embryo transfer group, all embryos will be cultured to D5 or D6. 1 blastocysts of the best quality will be transferred in fresh cycle on D5 or D6 after oocyte retrieval (D5 embryo will be the prior choice). The surplus embryos, if any, will be vitrified for future FET in case the fresh cycle does not result in a live birth. If a patient is at a high risk of OHSS, all embryos on D5 or D6 can be cryopreserved with vitrification for patient's safety. The FET cycle will be initiated on the second menstrual cycle after oocyte retrieval.
  Interventions: Procedure: blastocyst-stage embryo transfer
- cleavage-stage embryo transfer group (Experimental): For subjects assigned to the cleavage-stage (D2/3) embryo transfer group, 1 cleavage embryos of the best quality will be transferred in fresh cycle on Day 2/3 after oocyte retrieval. The surplus embryos, if any, will be vitrified for future FET if the fresh cycle does not result in a live birth. If a patient is at a high risk of OHSS, all embryos on Day 2/3 are allowed to be cryopreserved with vitrification for patient's safety. The FET cycle will be initiated on the second menstrual cycle after oocyte retrieval.
  Interventions: Procedure: cleavage-stage embryo transfer

INTERVENTIONS:
Procedure: blastocyst-stage embryo transfer — All the participants will receive a long GnRH-agonist, ultra-long GnRH-agonist, short GnRH-agonist or GnRH antagonist protocol in combination with recombinant FSH. HCG will be administered for final oocyte maturation. Patients will have a single blastocyst-stage embryos transferred. The outcomes of all the embryo transfers within 1 year after randomization will be followed up. Single embryo transfer (SET) is required for the first 3 embryo transfers within 1 year after randomization. For embryo transfers beyond the third within the 1 year, patients' treatment must follow their randomized allocation, and SET is no longer mandatory. Luteal phase support will be administered before embryo transfer. If pregnancy is confirmed, luteal phase support will be continued until 10 weeks of gestation. The follow up will be continued until 6 weeks after delivery.
  Arms: blastocyst-stage embryo transfer group
Procedure: cleavage-stage embryo transfer — All the participants will receive a long GnRH-agonist, ultra-long GnRH-agonist, short GnRH-agonist or GnRH antagonist protocol in combination with recombinant FSH. HCG will be administered for final oocyte maturation. Patients will have a single cleavage-stage embryos transferred. The outcomes of all the embryo transfers within 1 year after randomization will be followed up. Single embryo transfer (SET) is required for the first 3 embryo transfers within 1 year after randomization. For embryo transfers beyond the third within the 1 year, patients' treatment must follow their randomized allocation, and SET is no longer mandatory. Luteal phase support will be administered before embryo transfer. If pregnancy is confirmed, luteal phase support will be continued until 10 weeks of gestation. The follow up will be continued until 6 weeks after delivery.
  Arms: cleavage-stage embryo transfer group

SUMMARY:
The aim of this RCT is to compare differences in the efficacy and safety between cleavage-stage embryo transfer and blastocyst-stage embryo transfer in IVF/ICSI treatment cycle, taking into account of subsequent vitrified embryo transfers. Subjects with 3 or more transferrable cleavage embryos will be randomized to the cleavage-stage or blastocyst-stage embryos transfer group. The primary outcome is cumulative live birth rate (CLBR) per patient until the first live birth from one initiated oocyte retrieval cycle, calculated using outcomes from the first three embryo transfers within 1 year after randomization.

DETAILED DESCRIPTION:
This is a multicenter, randomized clinical trial comparing the efficacy and safety between cleavage-stage embryo transfer and blastocyst-stage embryo transfer in IVF/ICSI treatment cycle, taking into account of subsequent vitrified embryo transfers.Randomization will be performed on day 2/3 after oocyte retrieval, when at least 3 embryos are achieved. Patients in group A will have 1 cleavage-stage embryo transferred. Patients in group B will have 1 blastocyst-stage embryo transferred. The outcomes from all the embryo transfers within 1 year after randomization will be followed up. If a pregnancy/live birth is not achieved, single embryo transfer is required for the first 3 embryo transfers within 1 year after randomization. For embryo transfers beyond the third within the 1 year, patient's treatment must follow their randomized allocation, and SET is no longer mandatory. The follow-up period is 2 years from the day of randomization.Due to the COVID-19 pandemic, the participants who were unable to undergo the embryo transfers in 1 year of randomization will have 3 months extension for frozen embryo transfer. The follow-up for these participants will be extended for 3 months as well.

ELIGIBILITY:
Inclusion criteria:

1. Women aged ≥20 and ≤40 years.
2. Women with the number of transferrable cleavage embryos ≥ 3;
3. Women undergoing their first or second cycle of IVF or ICSI.

Exclusion criteria

1. Women who have been diagnosed with uterine abnormalities (confirmed by three-dimensional ultrasonography or hysteroscopy), including malformed uterus (uterus unicornis, septate uterus or duplex uterus), submucous myoma, or intrauterine adhesion
2. Women who plan to undergo In Vitro Maturation (IVM);
3. Women who plan to undergo Preimplantation Genetic Diagnosis (PGD) /Preimplantation Genetic Screening (PGS).
4. Women who have Women who have hydrosalpinx visible on ultrasound.
5. Women who have experienced recurrent spontaneous abortions, defined as 2 or more previous pregnancy losses.
6. Women who have been developed a "freeze-all" treatment plan for purpose of subsequent surgery, such as salpingectomy due to hydrosalpinx after oocytes retrieval.
7. Women with contraindications to assisted reproductive technology and/or pregnancy, such as uncontrolled hypertension, symptomatic heart diseases, uncontrolled diabetes, undiagnosed liver disease or dysfunction (based on serum liver enzyme test results), undiagnosed renal disease or abnormal renal function, severe anemia, history of deep venous thrombosis, pulmonary embolus or cerebrovascular accident, history of or suspicious for cancer, undiagnosed vaginal bleeding.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 992 (Actual)
Dates: Start 2018-09-29 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
cumulative live birth rate | 30 months
  Cumulative live birth rate (CLBR) is defined the first live birth per patient from one initiated oocyte retrieval cycle(Calculated using outcomes from the first three embryo transfers within 1 year after randomization). Live birth is defined as delivery of any neonate ≥24 weeks gestation with heart beat and breath.

SECONDARY OUTCOMES:
biochemical pregnancy rate | 30 months
  Biochemical pregnancy is defined as a serum β-HCG level of at least 25 IU/L 14 days after embryo transfer.
clinical pregnancy rate | 30 months
  Clinical pregnancy is defined by the presence of intrauterine gestation sacs at 30-35 days after embryo transfer.
ongoing pregnancy rate | 30 months
  Ongoing pregnancy is defined as a viable pregnancy at 12 weeks gestation.
Pregnancy loss rate | 30 months
  Pregnancy loss is defined as a pregnancy that results in a spontaneous abortion or therapeutic abortion that occurred throughout pregnancy.
moderate or severe OHSS rate | 12 months
  Number of patients with moderate or severe OHSS/ number of COS cycles.
ectopic pregnancy | 24 months
  diagnosed by ultrasound examination or laparoscopic surgery visualizing more than or equal to 1 gestational sacs outside the uterus or by abnormally increasing serum hCG level without sonographic visualization and the absence of chorionic villi inside the uterus after uterine curettage, which was treated by methotrexate.
sex ratio | 30 months
  the ratio of males to females in the newborns
multiple pregnancy | 30 months
  Number of multiple pregnancies / number of clinical pregnancies.
incidence of obstetric and perinatal complications | 30 months
  Number of pregnancies with complications / number of pregnancies; ;number of live births with neonatal complications / number of live births
congenital anomalies | 30 months
  structural or functional anomalies that occur during intrauterine life and can be identified prenatally, at birth or later in life.
implantation rate | 30 months
  the number of gestational sacs detected with sonography at 6 weeks of pregnancy/the number of embryos transferred
Birth weight | 30 months
  Weight of newborns at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Jiayin Liu, MD &PhD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Zi-Jiang Chen, MD &PhD, Principal Investigator — Center for Reproductive Medicine, affiliated to Shandong University
Locations (11):
- China (11):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Shengjing Hospital of China Medical University, Shenyang, Dongbei
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangxi Maternal and Child Health Hospital, Nanning, Guangxi
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Clinical Center of Reproductive Medicine at the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Center for Reproductive Medicine, Shandong Provincial Hospital Affiliated to Shandong University, Jinan, Shandong
  - Renji Hospital affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Suzhou Municipal Hospital, Suzhou, Suzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma X, Wang J, Shi Y, Tan J, Guan Y, Sun Y, Zhang B, Zhao J, Liu J, Cao Y, Li H, Zhang C, Chen F, Yi H, Wang Z, Xin X, Kong P, Lu Y, Huang L, Yuan Y, Liu H, Li C, Mol BWJ, Hu Z, Zhang H, Chen ZJ, Liu J. Effect of single blastocyst-stage versus single cleavage-stage embryo transfer on cumulative live births in women with good prognosis undergoing in vitro fertilization: Multicenter Randomized Controlled Trial. Nat Commun. 2024 Sep 5;15(1):7747. doi: 10.1038/s41467-024-52008-y. PMID 39237545